CLINICAL TRIAL: NCT03406247
Title: Adjuvant Immunotherapy After Salvage Surgery in Head and Neck Squamous Cell Carcinoma : Phase 2 Trial Evaluating the Efficacy and the Toxicity of Nivolumab Alone, and of the Combination Nivolumab and Ipilimumab
Brief Title: Adjuvant Immunotherapy After Salvage Surgery in Head and Neck Squamous Cell Carcinoma
Acronym: ADJORL1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-516810-39-00; 2017/2536 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental): Patients in cohorts 1 and 1bis will be administered Nivolumab 240 mg every 2 weeks during 3 first months and then 480 mg every 4 weeks during 3 months
  Interventions: Drug: Nivolumab
- Nivolumab + Ipilimumab (Experimental): Patients in cohorts 2 and 2bis will be administered
  * nivolumab 240 mg every 2 weeks during 6 months
  * ipilimumab 1mg/kg IV every 6 weeks during 6 months
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Patients in cohorts 1 and 1bis will be administered Nivolumab 240 mg every 2 weeks during 3 first months and then 480 mg every 4 weeks during 3 months Patients in cohorts 2 and 2bis will be administered
  - nivolumab 240 mg every 2 weeks during 6 months
Drug: Ipilimumab — Patients in cohorts 2 and 2bis will be administered
  - ipilimumab 1mg/kg IV every 6 weeks during 6 months
  Arms: Nivolumab + Ipilimumab

SUMMARY:
Two randomized trials of reirradiation after salvage surgery have been conducted by the GETTEC and GORTEC collaborative groups, both members of the French HN Intergroup: The first trial compared reirradiation and a "wait and see attitude" and was published in 2008 [1]. The second trial compared two modalities of reirradiation. Our hypothesis is that adjuvant treatment with immunotherapy will lead to a DFS similar to that observed in previous trials of post-operative reirradiation with possibly lower toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence or second primary of HNSCC in a previously irradiated area at a dose ≥ 50 Gys
* HNSCC of oral cavity, oro and hypopharynx, larynx only if extralaryngeal spread (rT4), isolated nodal recurrence
* Patient who has received salvage surgery with curative intent and macroscopic complete resection:
* for cohorts 1 and 2: similarly to inclusion criteria of previous reirradiation trials, more than 6 months between radiotherapy and salvage surgery
* for cohorts 1bis and 2bis: less than 6 months between radiotherapy and salvage surgery
* Recurrence of bad prognosis justifying an adjuvant treatment:
* clinically infiltrative recurrence or second primary; or nodal recurrence upper or equal to 3 cm, or association of local and nodal recurrence;
* superficial recurrence, but histologic gravity signs on surgical specimen indicating a high risk of recurrence after salvage surgery (histologic involvement of surgical margins or margins less than 3mm, perineural spread or vascular emboli, multiples invaded nodes). Nodal recurrence without tumor recurrence and inferior to 3cm, but with capsular rupture at histologic examination.
* Sufficient healing for beginning adjuvant treatment within 8 weeks (+/- 2 weeks) of salvage surgery
* No distant metastases, confirmed by CT or PET scan
* Male and female between 18 and 75 years (included)
* ECOG 0 or 1
* Immunosuppressive doses of systemic medication, such as steroids or absorbed topical steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before study drug administration
* Screening laboratory values must meet the following criteria (using CTCAE v4) and should be obtained within 14 days to the administration of the first study treatment.: WBC > 2,000/μL. Polynuclear neutrophils >1.5 x 10^9/L. Platelets > 75 x 10^9/L. Hemoglobin > 8.0 g/dL. ALAT/ASAT< 3.0 x ULN. Bilirubin < 1.5 x ULN (except Gilbert Syndrome

  : < 3.0 mg/dL). Creatinine clearance > 40 mL/min (measured or calculated by Cockroft and Gault formula) or serum creatinine < 2.0 x ULN
* Women of childbearing potential must have a negative serum β-HCG pregnancy test within 24 hours prior to the administration of the first study treatment.
* Sexually active women of childbearing potential must agree to use a highly effective method of contraception or to abstain from sexual activity during the study and for at least 5 months after the last study treatment administration. Sexually active males patients must agree to use condom during the study and for at least 7 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception.
* Women who are breastfeeding should discontinue nursing prior to the first dose of study drug and until 5 months after the last dose.
* Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Recurrent or metastatic carcinoma of the nasopharynx, squamous cell carcinoma that originated from the skin and salivary gland, or nonsquamous histologies (eg, mucosal melanoma).
* Recurrence or second primary of HNSCC in a non previously irradiated area, or at a dose < 50 Gys
* Macroscopic incomplete surgery (no debulking allowed)
* Superficial recurrence without nodal recurrence, and without histologic gravity signs (histologic involvement of surgical margins, perineural spread)
* Nodal recurrence less than 3 cm, without local recurrence and without capsular rupture at histologic examination
* Serious medical adverse conditions, such as severe cardiac and/or pneumologic and/or liver dysfunction. Non exhaustive list, to be appreciated in each center
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients with positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
* Patients with positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Patients having received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Patients receiving anti-cancer therapies must be discontinued at least 4 weeks prior to administration of study drug. Palliative, focal radiation therapy, and immunosuppressive doses of systemic corticosteroids, except replacement organotherapy (hydrocortisone and fludrocortisone), must be discontinued at least 2 weeks before administration of study drug. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (NCI CTCAE version 4) or to baseline or stabilized before administration of study drug. Subjects with toxicities attributed to systemic prior anticancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll.
* Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 4 weeks prior to study drug. The use of the inactivated seasonal influenza vaccine (Fluzone®) is allowed.Known or underlying medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events.
* Patients requiring concomitant treatment with therapeutic doses of anticoagulants will not be eligible for this clinical trial. Patients treated with low dose of anticoagulants for thrombo-embolic events prophylaxis are allowed.
* History of auto immune, immune mediated inflammatory disease including but not limited to colitis, pneumonitis, hepatitis, nephritis, inflammatory of skin, SNC, eyes, glands producing hormones
* Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
* History of severe hypersensitivity reaction to any monoclonal antibody
* History of allergy to study drugs components
* Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial
* Pregnancy or breastfeeding
* Psychological, familial or social factor incompatible with informed consent, and regular follow-up.
* Previous allogenic stem cell transplant or patients recipient of solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Two Years Disease Free Survival | Two years
  defined as the time from the beginning of the immunotherapy and the first locoregional or distant recurrence, or death from any cause, in cohorts 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Alix MARHIC, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided